



## Master Statistical Analysis Plan Checklist for Investigator Initiated Trials

A Two Arm Safety Study of Regorafenib before or after SIR-Spheres® Microspheres (90Y) for the Treatment of Patients with Refractory Metastatic Colorectal Cancer and Liver Metastases

Sponsor: Sarah Cannon Development Innovations

(Innovations)

Study Drug: SIR-Spheres® Microspheres

Protocol Number: GI 189

Prepared By: Innovations




REFERENCE SOP: CDS-0102

## Statistical Analysis Plan Checklist for Investigator Initiated Trials History of Changes

This document has undergone the following changes:

| Version Number | Version Date | Description of Changes |
|----------------|--------------|------------------------|
| 1.0 | 22MAY2018 | Original document |

Version Draft 1.0, 22 MAY 2018 





| 1.1 Objectives | |
|---|---|
| Primary Objective: | To evaluate the safety of two treatment cohorts combining regorafenib and SIR-Spheres microspheres (SIR-Spheres) radioemoblization in patients with refractory metastatic colorectal cancer (mCRC) with liver metastasis. |
| Secondary Objectives: | To evaluate the overall response rate (ORR), progression-free survival (PFS), and overall survival (OS) of patients with refractory mCRC when treated with combination SIR-Spheres and regorafenib in the two sequencing cohorts. |
| 1.2 Study Design | |
| Study Type | <ul><li>☑ Non-Randomized</li><li>☐ Randomized (Allocation Ratio: )</li></ul> |
| Details | This is an open-label study comparing the safety of two treatment cohorts in which radioembolization will be administered using the device SIR-Spheres microspheres (90Y resin microspheres) in combination with regorafenib to patients with mCRC with liver metastases. The two treatment cohorts will be evaluated for safety, ORR, PFS, and OS. Twenty-five patients will be treated in each cohort. The first cohort will complete enrollment before the second cohort opens. There will be no randomization or blinding. Blood samples will be collected from all patients prior to the hepatic angiogram and 99mTc MAA lung shunt scan, on Day 8 after SIR-Spheres treatment, and Day 30 (predose) after SIR-Spheres treatment (see Section 5.1). Expressions of cytokines and proteins will be measured to explore potential biomarkers that may correlate with clinical outcome. |
| 1.3.2 Randomization | |
| 1.3.2 Randomization Randomization Type: | ☐ Open-Label ☐ Single Blind ☐ Double-Blind |
| | ☑ Open-Label ☐ Single Blind ☐ Double-Blind |
| Randomization Type: | <ul> <li>☑ Open-Label ☐ Single Blind ☐ Double-Blind</li> <li>☐ Cohort Review / Dose Escalation</li> <li>☑ Safety Review</li> <li>☐ Interim Efficacy/Safety Analysis</li> <li>☐ Independent DMC/DSMB</li> <li>☐ Annual Report / Investigator Brochure (IB)</li> <li>☑ Abstract / Scientific Presentation (Oral/Poster)</li> </ul> |
| Randomization Type: 1.4 Timing of Analysis | ☐ Cohort Review / Dose Escalation ☐ Safety Review ☐ Interim Efficacy/Safety Analysis ☐ Independent DMC/DSMB ☐ Annual Report / Investigator Brochure (IB) |
| Randomization Type: 1.4 Timing of Analysis Planned Interim Analysis | ☐ Cohort Review / Dose Escalation ☐ Safety Review ☐ Interim Efficacy/Safety Analysis ☐ Independent DMC/DSMB ☐ Annual Report / Investigator Brochure (IB) ☐ Abstract / Scientific Presentation (Oral/Poster) |
| Randomization Type: 1.4 Timing of Analysis Planned Interim Analysis Final Analysis | ☐ Cohort Review / Dose Escalation ☐ Safety Review ☐ Interim Efficacy/Safety Analysis ☐ Independent DMC/DSMB ☐ Annual Report / Investigator Brochure (IB) ☐ Abstract / Scientific Presentation (Oral/Poster) |
| Randomization Type: 1.4 Timing of Analysis Planned Interim Analysis Final Analysis 1.5 Responsibilities | □ Cohort Review / Dose Escalation □ Safety Review □ Interim Efficacy/Safety Analysis □ Independent DMC/DSMB □ Annual Report / Investigator Brochure (IB) □ Abstract / Scientific Presentation (Oral/Poster) 6 months after last patient has been recruited into study Development of SAP and shells |

Version Draft 1.0, 22 MAY 2018 





REFERENCE SOP: CDS-0102

| 1.6 Analysis Software | |
|----------------------------|--------------------------|
| Main statistical analysis: | SAS Version 9.3 or above |
| Other analysis software: | None |

| 1.7 Coding | |
|---|---|
| <ul><li>☑ Adverse Events</li><li>☐ Medical History</li></ul> | <ul> <li>✓ MedDRA:</li></ul> |
| <ul><li>☐ Concomitant Medication</li><li>☐ Prior Therapy</li><li>☐ Subsequent/Further</li><li>Therapy</li></ul> | <ul> <li>☑ WHO-Drug: ☐ Version</li> <li>☑ Most current release and update coding with new major releases</li> </ul> |
| 3 Analysis Population | |
| Intent-To-Treat (ITT) Population definition: | <ul> <li>☑ All patients who have started treatment in the study</li> <li>☐ All patients who have been randomized in the study, regardless of whether they have received any treatment or not</li> <li>☐ All patients who have been randomized and have started treatment in the study</li> <li>☐ Other definition, specify:</li> </ul> |
| Per Protocol (PP) Population to be used in analysis: | ☐ Yes ☐ No If yes, please specify the criteria for exclusion from the PP population: |
| Safety (SAF) Population definition | <ul> <li>☑ All patients who have started treatment in the study. Patients will be analyzed according to the actual treatment they have received.</li> <li>☐ Other definition, specify:</li> </ul> |
| Other Analysis Population definition: | N/A |
| 4 Baseline Value Definitions | |
| | Last value prior to first date of study drug treatment |
| 5/6 Efficacy | |
| Response Criteria Used: | ☐ RECIST 1.0 ☐ RECIST 1.1 ☐ Cheson 2007 ☐ Modified RECIST – specify: ☐ Other criteria, Specify: |

Version Draft 1.0, 22 MAY 2018 





REFERENCE SOP: CDS-0102

| Efficacy Assessment Timepoints: | Assessed during treatment at week 6 and week 12. Patients continuing treatment after week 12 will be assessed at 8 week intervals. Patients with progressive disease (PD), unacceptable toxicity, or who withdraw consent will be removed from the study. | | | | |
|---|---|---|---|---|---|
| | Patients will be assessed at end of treatment visit | | | | |
| | During follow-up, patients will be assessed every 3 months up to 6 months. | | | | |
| Efficacy Endpoints: | | | | | |
| | | Endpoint | Primary Analysis<br>Population | Other Anal<br>Population | |
| | Primary | Overall Response<br>Rate (ORR) | ITT Population | | |
| | Secondary | Progression-Free<br>Survival (PFS) | ITT Population | | |
| | | Overall Survival (OS) | | | |
| <b>Definition of Terms:</b> | | | | | |
| ⊠ Response | ☐ Complete F | <ul> <li>☐ Complete Response + Partial Response as best observed response</li> <li>☑ Complete Response + Partial Response, confirmed with 4 weeks apart.</li> <li>☐ Other criteria, specify:</li> </ul> | | | |
| ☐ Clinical Benefit | response Complete F Stable Dise | <ul> <li>☐ Complete Response + Partial Response + Stable Disease as best observed response</li> <li>☐ Complete Response + Partial Response (confirmed with stable Disease (at least weeks from start of treatment)</li> <li>☐ Other criteria, specify:</li> </ul> | | | |
| ☑ Progression | As defined in A | As defined in Appendix C of the protocol. | | | |
| ☐ Subsequent Therapy | | | | | |
| ☐ Treatment Failure | | | | | |
| Definition of Endpoints: | End Date (spe | Start Date: Date of Randomization Date of First Treatment End Date (specify for all pertinent endpoints): Overall Survival: Event = Death | | | |
| | | Situation | Date of Event of | or Censoring | Outcome |
| | Death | | Date of death | | Event |
| | Alive on date | of data cutoff | Date last known | າ alive | Censored |
| | Alive before date of data cutoff, but status unknown on date of data cutoff (e.g. lost to follow-up) Ce | | Censored | | |

Version Draft 1.0, 22 MAY 2018 



| | Progression-Free Survival: Event = Progression of | or Death | |
|---|---|---|---|
| | Situation | Date of Event or Censoring | Outcome |
| | No baseline assessment | Date of first treatment | Censored |
| | Progression documented between scheduled visits | First date of evaluated overall response = PD | Event |
| | No progression | Date of last evaluable tumor assessment | Censored |
| | Treatment discontinuation for adverse event or other reason | Date of last evaluable tumor assessment | Censored |
| | Death before first PD assessment | Date of death | Event |
| | Death before the next scheduled tumor assessment | Date of death | Event |
| | Death after one missed tumor assessment but before second missed tumor assessment | Date of death | Event |
| | Death after two or more missed tumor assessment | Date of last evaluable tumor assessment | Censored |
| ☑ Overall Response Rate (ORR) | Default: Estimates of rates in each treatment | arm | |
| ☐ Disease Control Rate (DCR) | <ul><li>☑ Difference in rates &amp; 95% confidence inte</li><li>☑ p-value, specify statistical test:</li></ul> | erval between treatment arm | S |
| ☐ Clinical Benefit Rate (CBR) | — p-value, specify statistical test. | | |
| ☐ Early Progression Rate (EPR) | | | |
| ☐ Time To Progression (TTP) | Default: Estimates of medians in each treatm | | |
| ☑ Progression-Free Survival (PFS) | ☐ Other quartiles or percentages of survival required, specify: probability evaluates 6 month intervals | | |
| Overall Survival (OS) | ☐ Hazard ratio & 95% confidence interval b | etween treatment arms, uns | ıratıneti |
| ☐ Duration of Response | ☐ Hazard ratio & 95% confidence interval between treatment arms, stratified (specify stratification factor(s)): | | |
| ☐ Duration of Stable Disease | p-value, specify statistical test: | | |
| ☐ Time To Treatment Failure (TTF) | | | |
| Other, Specify: | | | |
| 7 Safety | | | |
| Adverse Events | Definition of Treatment-Emergent Adverse E starts or worsens after the start of the first do last dose. | | |
| Laboratory Data | Data will be summarized by: | | |
| | | eters, and H/L for non-CTCA | E-Gradable |

Version Draft 1.0, 22 MAY 2018 




REFERENCE SOP: CDS-0102

| H/L for all lab parameters |
|----------------------------|

## Tier 1 Study - Tables, Figures & Listings

| Standard TFLs | | | |
|---|---|---|---|
| Table No | Description | Variables/Analyses To Be Included | Subgroup Analyses |
| Table 1 | Summary of Demographics and Disease Characteristics | <ul> <li>☒ Age: Median, Min, Max</li> <li>☐ Age Group:</li> <li>☒ Sex</li> <li>☒ Race</li> <li>☒ ECOG</li> <li>☒ Other, specify: Primary diagnosis, KRAS, BRAF</li> </ul> | Safety Analysis Set |
| Table 2 | Summary of Metastatic Involvement at study entry | ☐ Histology ☐ Disease Staging ☐ Time from Diagnosis ☐ Other, specify: sites of metastatic involvement (count and percent of patients per involved site) | Safety Analysis Set |
| Table 3 | Summary of Regorafenib Exposure and Treatment Modifications | Treatment duration, number of patients with each treatment modification, reasons for dose modifications | Safety Analysis Set |
| Table 4 | Summary of SIR-Spheres Exposure | Activity delivered to liver (mCi), lung shunt fraction, total tumor volume (mL): number of patients, Mean, SD, Median, Min, Max | Safety Analysis Set |
| | | Treatment planning (left, right, whole): number and percent of patients | |
| Table 4 | Summary of Treatment Discontinuations | Number of patients with treatment discontinuation, reasons for treatment discontinuation | Safety Analysis Set |
| Table 5 | Summary of Best Overall Response | Best overall response: Complete response (CR), Partial response (PR), Stable disease (SD), progressive disease (PD), not evaluable (NE) | ITT Population/Efficacy<br>Analysis Set |
| | | Objective response rate (ORR) (CR + PR): ORR, 95% Confidence interval | |
| | | CR and PR confirmed | |
| Table 6 | Summary of Progression-Free Survival | Kaplan-Meier | ITT Population/Efficacy |
| | | Number of patients with events,<br>Number of patients censored, Median,<br>25 <sup>th</sup> and 75 <sup>th</sup> percentiles for progression<br>free survival [months (95% CI)] | Analysis Set |
| | | Probability of events evaluated in 6 month intervals | |
| Table 7 | Summary of Overall Survival | Kaplan-Meier | ITT Population/Efficacy<br>Analysis Set |

Version Draft 1.0, 22 MAY 2018 






REFERENCE SOP: CDS-0102

| Standard TFLs | | | |
|---|---|---|---|
| Table No | Description | Variables/Analyses To Be Included | Subgroup Analyses |
| | | Number of patients with events,<br>Number of patients censored, Median,<br>25 <sup>th</sup> and 75 <sup>th</sup> percentiles for overall<br>survival [months (95% CI)]<br>Probability of events evaluated in 6<br>month intervals | |
| Table 8 | Summary of Treatment-Related<br>Adverse Events | Sarah Cannon/Modified CTCAE coding By CTCAE grade | Safety Analysis Set |

| Figure<br>No | Description | Variables/Analyses To Be Included | Subgroup Analyses |
|---|---|---|---|
| Figure 1 | Progression-Free Survival | Timescale to be used on horizontal axis: ☐ Day ☐ Week ☐ Month ☐ Year | ITT Population/Efficacy<br>Analysis Set |
| Figure 2 | Overall Survival | Timescale to be used on horizontal axis: ☐ Day ☐ Week ☐ Month ☐ Year | ITT Population/Efficacy<br>Analysis Set |

Version Draft 1.0, 22 MAY 2018 